CLINICAL TRIAL: NCT06072456
Title: Comparison of Vaginal Axis on MRI in Alternative Apical Prolapse Surgeries to Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, fatih sahin, Principal Investigator, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-10840098-772.02-4704
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; apical prolapse; pectopexy; sacrospinous ligament fixation; Lateral suspension
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- lateral suspension (Experimental): Suspending the cervix to the bilateral abdominal wall through subperitoneal tunnels may properly mimic cardinal ligament and restore the normal vaginal axis. Preoperative and postoperative MRI results were evaluated
  Interventions: Procedure: laparoscopic lateral suspension
- pectopexy (Experimental): The cervix or vaginal cuff was suspended by the Cooper ligament.Preoperative and postoperative MRI results were evaluated
  Interventions: Procedure: laparoscopic pectopexy
- sacrospinous ligament fixation (Experimental): vaginal cuff/uterus was sutured to the unilateral sacrospinous ligament.Preoperative and postoperative MRI results were evaluated
  Interventions: Procedure: Sacrospinous ligament fixation
- hysterectomized patients (No Intervention): Vaginal axis MRI of women who have previously been hysterectomized and who do not have apical prolapse
- Nulliparous women (No Intervention): MRI of nulliparous women was evaluated for vaginal axis.

INTERVENTIONS:
Procedure: laparoscopic lateral suspension — Lateral suspension involves the lateral attachment or suspension of vaginal tissue to a stable structure, often using mesh or sutures, to provide support and stability to the pelvic organs. Control groups consist of hysterectomized women without cuff prolapse and nulliparous women.
  Arms: lateral suspension
Procedure: laparoscopic pectopexy — Pectopexy involves attaching or suspending the vaginal vault to the pectineal ligament, which is a strong ligament in the pelvis. Control groups consist of hysterectomized women without cuff prolapse and nulliparous women.
  Arms: pectopexy
Procedure: Sacrospinous ligament fixation — Sacrospinous ligament fixation entails the attachment or fixation of the vaginal vault to the sacrospinous ligament, which is a strong fibrous band located in the pelvis
  Arms: sacrospinous ligament fixation

SUMMARY:
Sacrocolpopexy remains the preeminent modality in addressing apical prolapse surgically. Nevertheless, amplified morbidity rates within cohorts characterized by obesity and advanced age constrain the advantages conferred by the procedure. Recent years have witnessed a proliferation of inquiries appraising the efficacy of laparoscopic lateral suspension, pectopexy, and sacrospinous ligament fixation interventions, which have, over time, garnered extensive clinical application, in relation to recurrence rates. A multitude of investigations have been undertaken to delineate the optimal vaginal axis. In the present investigation, we have delineated a research protocol aimed at scrutinizing these alternative surgical modalities with regard to their impact on the vaginal axis.

DETAILED DESCRIPTION:
The study objective pertains to the assessment of vaginal axis in patients undergoing apical prolapse surgery, whether they have undergone hysterectomy or not. The investigation is designed to test the null hypothesis by means of a comparative analysis of preoperative and postoperative Magnetic Resonance Imaging images capturing the vaginal axis. This examination will be conducted on patients slated to receive lateral mesh suspension, pectopexy, and sacrospinous ligament fixation procedures for the correction of apical prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Female with genital prolapse

Exclusion Criteria:

* Patients who had pouch of Douglas obliteration
* Patients with enterocele
* Patients who have any congenital or acquired anatomic and reproductive anomaly

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Vaginal axis | at 4th months after the operation
  From the images obtained in the sagittal plane, the vagina, which will be observed as a high signal intensity linear structure in T2A images, and the levator plate extending as a flow-signal intensity flat structure in T1A images, will be evaluated.
Vaginal distances | at 4th months after the operation
  The distance between the posterior vaginal fornix and the midpoint of the anterior side of the 2nd vertebra will be measured in the mid-sagittal plane (PF-S2). The distance between the right spina ischiadica and right vaginal fornix (RSI-RF), and, the distance between the left spina ischiadica and left vaginal fornix (LSI-LF) will be measured on T2A images acquired in the axial plane.

SECONDARY OUTCOMES:
Prolapse symptoms, Colorectal-Anal Impact Questionnaire | at 4th months after the operation
  The Pelvic Floor Impact Questionnaire-Short Form 7 (PFIQ-7) consists of three scales of seven questions, each taken from the Urinary Incontinence Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The three scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300) describes the impact on day to day activities. It is useful to determine changes in symptom-severity over time and before and after treatments
Prolapse symptoms | at 4th months after the operation
  The Pelvic Floor Distress Inventory-Short Form 20 (PFDI-20) measures both pelvic floor symptoms and the degree of bother and distress associated with those symptoms. The PFDI-20 includes 20 questions and three scales. Each of the three scales is scored from 0 (least distress) to 100 (greatest distress), again with an overall score ranging from 0-300 and higher scores indicating lower quality of life. The three scales include questions taken from the Urogenital Distress Inventory-6 questions, the Pelvic Organ Prolapse Distress Inventory-6 questions, and the Colorectal-Anal Distress Inventory-8 questions.
Urinary Symptoms | at 4th months after the operation
  Validated scales were applied for this purpose, including the urogenital distress inventory-6 (UDI-6), which is a shortened version of a condition-specific quality of life instrument. The UDI-6 is frequently used due to its feasibility and is validated at level A according to the International Continence Society (ICI) grading system. The UDI-6 scale includes six items that assess various aspects of urinary symptoms and their impact on daily life. These items include: 1) Frequent urination, 2) Leakage related to the feeling of urgency, 3) Leakage related to activity, 4) Coughing or sneezing small amounts of leakage (drops), 5) Difficulty emptying the bladder, and 6) Pain or discomfort in the lower abdominal or genital area. Higher scores on the UDI-6 indicate a higher level of disability in these areas.
Postoperative de novo dyspareunia | at 4th months after the operation
  Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) Postoperative de novo dyspareunia assessed by the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) with main focus on Question 5, which represents how the participant feels about her sex life (I feel frustrated by my sex life/I feel sexually inferior because of my incontinence and/or prolapse/I feel angry because of the impact that incontinence and/or prolapse has on my sex life)
Sexual functions | at 4th months after the operation
  The Female Sexual Function Index (FSFI) evaluates sexual functioning in women and comprises of 19 questions with different answer choice scales referring the sexual life in the previous 4 weeks. The answer choices in the FSFI carry a number of points and are summed to obtain six domain scores and an overall score. For the latter, there is a threshold at 26.55 which means that all values below are classed as indicating female sexual dysfunction (FSD). The domain scores are obtained as the sum of points attributed to questions in that domain multiplied by the domain factor.
Quality of life measures | at 4th months after the operation
  General health Short Form Health Survey (SF-12) Form includes two questions concerning physical functioning; two questions on role limitations due to physical health problems; one question on bodily pain; one question on general health perceptions; one question on vitality (energy/fatigue); one question on social functioning; two questions on role limitations due to emotional problems; and two questions on general mental health (psychological distress and psychological well-being
Patient Global Impression of Improvement (PGI-I) | at 4th months after the operation
  Patient Global Impression of Improvement (PGI-I). A low score on the PGI-I indicates an overall improvement in a woman's perception of her condition after treatment (PGI-I score of 1 or 2 = very much better and much better, respectively

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cemil Taşcıoğlu Hospital, Istanbul
  - Prof.Dr.Cemil Taşcıoğlu Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Senturk MB, Kilicci C, Aydin S, Polat M, Abide Yayla C, Karateke A. Vaginal axis on MRI after unilateral and bilateral sacral hysteropexy: a controlled study. J Obstet Gynaecol. 2018 Jan;38(1):115-120. doi: 10.1080/01443615.2017.1336754. Epub 2017 Aug 17. PMID 28816554
- [Result] Pulatoglu C, Yassa M, Turan G, Turkyilmaz D, Dogan O. Vaginal axis on MRI after laparoscopic lateral mesh suspension surgery: a controlled study. Int Urogynecol J. 2021 Apr;32(4):851-858. doi: 10.1007/s00192-020-04596-8. Epub 2020 Nov 11. PMID 33175232